CLINICAL TRIAL: NCT02505152
Title: Percutaneous Transhepatic Intrahepatic Portosystemic Shunt for Treatment of Portal Vein Occlusion With Symptomatic Portal Hypertension After Splenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zaibo Jiang, Department of Radiology, The Third Affiliated Hospital, Sun Yat-Sen University, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTIPSDORNO3HSYSU
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension, Portal; Portal Vein, Cavernous Transformation Of
Keywords: Hypertension, Portal; Portal Vein, Cavernous Transformation Of; Portosystemic shunt; Radiology, Interventional
MeSH Terms: conditions — Hypertension, Portal; Portal Vein, Cavernous Transformation Of

ARMS (1):
- Shunt (Experimental): Perform percutaneous transhepatic intrahepatic portosystemic shunt
  Interventions: Procedure: Percutaneous transhepatic intrahepatic portosystemic shunt

INTERVENTIONS:
Procedure: Percutaneous transhepatic intrahepatic portosystemic shunt — Under fluoroscopic guidance, portal vein(PV) was punctured with a 22-gauge Chiba needle. A 0.018-inch guidewire was advanced through the needle into PV lumen. The needle was exchanged and a 7-French sheath inserted over the wire. Then retrohepatic inferior vena cava(RIVC) or hepatic vein(HV) was punctured with a 20-gauge, 30-cm Chiba needle through sheath. Another 0.018-inch guidewire was advanced through the needle into right internal jugular vein and then snared out of body. A 0.035-inch, 260-cm stiff shaft wire was then introduced through the transjugular sheath and manipulated into main portal vein(MPV) and then into superior mesenteric vein(SMV). Afterward the PTIPS procedure was completed in the standard transjugular fashion.

SUMMARY:
To evaluate the values of percutaneous transhepatic intrahepatic portosystemic shunt for treatment of portal vein occlusion with symptomatic portal hypertension after splenectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with portal hypertension who have the history of splenectomy and have enough image information to confirm occlusion of portal vein

Exclusion Criteria:

* Patients with known severe dysfunction of heart, lung, brain, kidney and other vital organs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
No gastrointestinal rebleeding in 1 month after interventions | 1 month
  No gastrointestinal rebleeding in 1 month after interventions
Ascites disappear in 1 month after interventions | 1 month
  Ascites disappear in 1 month after interventions

SECONDARY OUTCOMES:
Whether the shunt is patent after interventions in 6 months | 6 months
  Patent shunt in 6 months after interventions proved by US or CT

CONTACTS AND LOCATIONS:
Overall Officials: Zaibo Jiang, MD., Study Chair — Sun Yat-sen University
Locations (1):
- Department of Radiology, Guangzhou, Guangdong, China